CLINICAL TRIAL: NCT03191825
Title: Testing the Efficacy of a Lapse Management System in an Online Smoking Cessation
Brief Title: Online Lapse Management Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Håvar Brendryen, Senior researcher, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFR 228158/H10
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Nicotine Dependence, Cigarettes
Keywords: online intervention; mHealth m-Health; eHealth e-Health; smoking cessation; lapse management; relapse prevention
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: All participants receive one out of three versions of a web-based smoking cessation program. Two of the versions includes a lapse management system that are based on a day-to-day logging of target behavior. In one version the logging is done on the web, while on the other version, logging is done by SMS-textmessages.
Masking Description: The recruitment procedure and the treatment is fully automated and delivered by web, e-mail and SMS-textmessages - i.e., the participant is not contacted by any care providers, investigators or assessors during recruitment or treatment - and data are collected by means of web-based questionnaires. However, non-responders to the questionnaires will be contacted by phone for telephone interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard web-application (Active Comparator): Endre: a digital smoking cessation counsellor
  Interventions: Other: Endre: a digital smoking cessation counsellor
- Web-based lapse management system (Experimental): Endre: a digital smoking cessation counsellor + Lapse management system triggered from web-page
  Interventions: Other: Endre: a digital smoking cessation counsellor; Other: Lapse management system triggered from web-page
- SMS & web-based lapse management system (Experimental): Endre: a digital smoking cessation counsellor + Lapse management system triggered by SMS-textmessage
  Interventions: Other: Endre: a digital smoking cessation counsellor; Other: Lapse management system triggered by SMS-textmessage

INTERVENTIONS:
Other: Endre: a digital smoking cessation counsellor — A comprehensive 25-session intervention delivered by web, e-mail and SMS-text messages. Sessions are released one each day for 18 days, and then every second day for 14 days. Intervention content is tailored based on user input and individual usage pattern. The intervention is described in detail in Holter, Johansen & Brendryen (2016). How a fully automated eHealth program simulates three therapeutic processes: A case study. Journal of Medical Internet Research 18 (6).
Other: Lapse management system triggered from web-page — The lapse management system is based on a day-to-day logging of the target behavior (smoking). This logging goes on for four weeks after an initial quit attempt. The current version of the system logs by asking the participant about their smoking status every time they log on to "Endre" (the digital smoking cessation counsellor). Participants that report a lapse is routed to a fully automated counselling session delivered by web.
  Arms: Web-based lapse management system
Other: Lapse management system triggered by SMS-textmessage — The lapse management system is based on a day-to-day logging of the target behavior (smoking). This logging goes on for four weeks after an initial quit attempt. The current version of the system logs by asking the participant about their smoking status in a textmessage (SMS) sent each evening. Participants that report a lapse, receives a new SMS with a link to a fully automated counselling session delivered by web.
  Arms: SMS & web-based lapse management system

SUMMARY:
The purpose of the trial is to test the adjunctive effect of adding a lapse management system to a best practices web- and mobile smoking cessation program.

DETAILED DESCRIPTION:
Background: Web- and mobile phone health behavior change interventions, including smoking cessation programs, offer great promise, but little is known about the components that may add to their effect.

Objectives: To assess tobacco abstinence associated with an adjunctive lapse management system combined with a best-practices web- and mobilephone based smoking cessation intervention. The investigators hypothesize that a program that includes the lapse management system will yield greater efficacy than a program that does not include such a component.

Methods: The investigators propose a 3-arm RCT with 1500 adult study participants that all receive a best practices web-based smoking cessation program designed for use on snart phones (web-app). Participants are randomized to either the web-app only, the web-app plus a web-based lapse management system, or web-app plus a SMS-based lapse management system.

The lapse management system will be based on the day-to-day logging of target behavior and providing just-in-time therapy to clients reporting a lapse. In the two versions of the lapse management system the logging of target behavior is done by asking a question about smoking status by web or SMS.

Measures: The primary outcome is 7-day point prevalence tobacco abstinence (as assessed at the 1- and 6-months follow-up). Potential predictors, moderators, and mediators of abstinence will also be examined.

Benefits: This protocol describes the first RCT that assesses the incremental efficacy of adding a lapse management system to an online smoking cessation intervention. These interventions constitute a cost-effective means to reach smokers who want to quit. By seeking to identify beneficial adjunctive mechanisms, their efficacy may be improved, which can make a substantial public health impact.

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* beeing a current smoker
* determined to or considering to quit smoking
* provide valid e-mail address
* provide valid norwegian cell phone number
* complete a baseline questionnaire
* complete a ten day run-in period (preparation phase)
* reporting an initial quit attempt ("yes, today I have quit smoking")

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
7 day point prevalence abstinence from cigarettes | measured at six months post cessation
  no tobacco smoking during the last seven days

SECONDARY OUTCOMES:
7 day point prevalence abstinence from cigarettes | measured at one month post cessation
  no tobacco smoking during the last seven days
7 day point prevalence abstinence from any nicotine products | measured at one month post cessation
  no use of products containing nicotine (smoking tobacco, snuff, e-cigarettes, nicotine replacement products etc) during the last seven days
7 day point prevalence abstinence from any nicotine products | measured at six months post cessation
  no use of products containing nicotine (smoking tobacco, snuff, e-cigarettes, nicotine replacement products etc) during the last seven days

OTHER OUTCOMES:
user engagement | during a one month timeframe after initial quit attempt
  number of completed sessions after initial quit attempt
number of lapse episodes after initial quit attempt | assessed one month after cessation day
  lapse episode = experiencing a temporary setback, i.e., smoking one or several cigarettes and then beeing abstinent again

CONTACTS AND LOCATIONS:
Overall Officials: Håvar Brendryen, PhD, Principal Investigator — University of Oslo
Locations (2):
- Department of Addictology, 1st Faculty of Medicine, Charles University, Prague, Czechia
- The Norwegian Centre for Addiction Research, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holter MT, Johansen A, Brendryen H. How a Fully Automated eHealth Program Simulates Three Therapeutic Processes: A Case Study. J Med Internet Res. 2016 Jun 28;18(6):e176. doi: 10.2196/jmir.5415. PMID 27354373
- See also: Official home page for PI at host institution — https://www.sv.uio.no/psi/english/people/aca/haavabre/index.html
- See also: PIs Google Schoolar Profile — https://scholar.google.no/citations?user=i3m0lqgAAAAJ&hl=en&oi=ao